CLINICAL TRIAL: NCT03859765
Title: Development and Pilot Testing of a Hybrid In Person and mHealth Coping Skills Training Intervention for Symptom Management and Daily Steps in Stem Cell Transplant Patients
Brief Title: In Person and mHealth Coping Skills Training for Symptom Management and Steps in Stem Cell Transplant Patients
Acronym: Symptoms-Steps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100321
Record Dates: First submitted 2019-02-12; First posted 2019-03-01 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2022-09

CONDITIONS: Stem Cell Transplant
Keywords: physical disability; pain; fatigue; distress; physical activity; coping; mHealth; cancer; symptom management
MeSH Terms: conditions — Pain; Fatigue; Motor Activity; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCT Symptoms and Steps (Experimental): HCT Symptoms and Steps participants will complete in-person (3) and video-conferencing (4) coping skills training and activity coaching sessions teaching cognitive behavioral coping skills to manage pain, fatigue, and distress and increase activity. Participants will be given a wireless activity tracker and a smartphone for accessing the study mobile app.
  Interventions: Behavioral: HCT Symptoms and Steps
- HCT Education (No Intervention): HCT Education participants will receive 1 brief in clinic session prior to discharge home providing education related to symptom management and physical activity, and a wireless activity tracker. HCT Education participants will also receive 6 brief phone calls upon return home.

INTERVENTIONS:
Behavioral: HCT Symptoms and Steps — HCT Symptoms and Steps will provide patients with cognitive behavioral coping skills training and activity coaching sessions to enhance their ability to manage symptoms that interfere with activity.
  Arms: HCT Symptoms and Steps

SUMMARY:
Hematopoietic stem cell transplant (HCT) is an aggressive treatment for life-threatening cancers. HCT improves survival, but most HCT patients experience significant physical disability, which is exacerbated by persistent symptoms. Pain, fatigue, and psychological distress are the most prevalent and debilitating symptoms. HCT patients experience a significant increase in disability as their pain, fatigue, and distress increase. This disability and symptom burden interferes with patients' ability to engage in recommended physical activity that can improve disability, symptoms, and other outcomes. Disability and symptoms also complicate an already challenging recovery course; HCT patients return home, often far from their medical team, are restricted from normal activities and socially isolated. These disability, symptom and activity challenges increase the risk for post-transplant complications and may compromise life expectancy. Teaching HCT patients to cope with symptoms and activity is critical to helping them increase activity and reduce disability. Cognitive behavioral coping skills training protocols can enhance HCT patients' ability to cope with symptoms (pain, fatigue, distress) that interfere with physical activity. However, the application of these protocols to HCT patients is limited by in person sessions, delivery of sessions in a medical center setting, and/or lack of tailoring to HCT patients' specific needs. Mobile health (mHealth) technologies can improve and extend intervention strategies to cope with symptoms and physical activity upon return home. Behavioral intervention strategies are needed to enable HCT patients to effectively cope with symptoms to improve their ability to engage in physical activity that can improve physical disability.

The investigators aim to develop and test a combined coping skills training and activity coaching protocol that: first, is feasible and acceptable, and second, improves physical disability, as well as pain, fatigue, distress, and physical activity in HCT patients. Specifically, the investigators will develop and test an in-person and mHealth HCT Coping Skills Training for Symptom Management and Daily Steps (HCT Symptoms and Steps) intervention protocol. To do this, the investigators will develop a mobile app, conduct focus groups, complete user testing, and conduct a small randomized controlled trial (RCT) to examine feasibility, acceptability, and outcome patterns suggesting intervention efficacy of the developed HCT Symptoms and Steps protocol. Following the development phase of the study (i.e., focus groups), the investigators will conduct user testing with 10 cancer patients who have undergone HCT; all 10 patients will receive the HCT Symptoms and Steps intervention. Next, the investigators will randomly assign 40 cancer participants who have undergone HCT and report pain, fatigue and stress to receive either HCT Symptoms and Steps or HCT Education. The investigators will test whether HCT Symptoms and Steps is feasible and acceptable to HCT patients, and improves physical disability, as well as other important outcomes. The investigators expect that HCT Symptoms and Steps will be feasible and acceptable to HCT patients and, compared to HCT Education, will be more likely to lead to improvements in physical disability, as well as pain, fatigue, distress, physical activity, and self-efficacy for symptom management.

The investigators' goal is to demonstrate the feasibility, acceptability, and positive impact of a hybrid in-person and mHealth coping skills training and activity coaching intervention that reduces physical disability by concurrently and synergistically decreasing symptom burden and increasing physical activity. This project has the potential to lead to future research that can redesign existing modes of behavioral intervention delivery, improve continuity and coordination of care, and ultimately enhance patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hematopoietic stem cell transplant due to oncological disease
* Clinical ratings of pain, fatigue and psychological distress
* Life expectancy of 12 or more months

Exclusion Criteria:

* Cognitive impairment
* Severe psychiatric condition
* Inability to converse in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

REFERENCES:
- [Derived] Kelleher SA, Fisher HM, Hyland K, Miller SN, Amaden G, Diachina A, Pittman AS, Winger JG, Sung A, Berchuck S, Samsa G, Somers TJ. Hybrid-delivered cognitive behavioral symptom management and activity coaching intervention for patients undergoing hematopoietic stem cell transplant: Findings from intervention development and a pilot randomized trial. J Psychosoc Oncol. 2023;41(5):539-557. doi: 10.1080/07347332.2022.2152519. Epub 2022 Dec 8. PMID 36476318

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HCT Symptoms and Steps | HCT Education
Started | 20 | 20
Completed | 17 | 18
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HCT Symptoms and Steps | HCT Education | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 14 | 25
  >=65 years | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.59 (11.04) | 58.5 (10.96) | 59.32 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 19 | 17 | 36
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Cancer Type [Count of Participants; unit: Participants]
  Lymphoma | 1 | 5 | 6
  Multiple Myeloma | 17 | 14 | 31
  Other | 2 | 1 | 3
First cancer or recurrence [Count of Participants; unit: Participants]
  First Cancer | 17 | 13 | 30
  Recurrence | 3 | 7 | 10
Time since diagnosis (months) [Mean (Standard Deviation); unit: Months] | 33.46 (65.08) | 18.86 (30.60) | 26.16 (50.73)
Number of participants receiving chemotherapy [Count of Participants; unit: Participants] | 7 | 8 | 15
Number of participants receiving anti-cancer drug [Count of Participants; unit: Participants] | 3 | 2 | 5
Time since transplant (days) [Mean (Standard Deviation); unit: Days] | 25.10 (44.30) | 14.20 (10.98) | 19.65 (32.33)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Number of Participants Accrued to the Study Within 16 Months
Description: Feasibility will be shown by meeting targeted study accrual (N=40) in the 16-month study period.
Time Frame: 16 months (additional year granted due to COVID-19).
Population: Total number screened
Measure: Count of Participants; unit: Participants
Groups:
- Screening: Potential participants who were screened prior to consent
Arm/Group | Screening
Number analyzed (Participants) | 123
Participants
  Number Ineligible | 28
  Number Eligible but Declined | 51
  Number Eligible but Unable to Consent | 4
  Number Accrued | 40

2. Primary Outcome: Number of Participants Who Adhere to at Least 80% of the Study Protocol
Description: A measure of feasibility.
Time Frame: approximately 20-24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HCT Symptoms and Steps | HCT Education
Number analyzed (Participants) | 20 | 20
Participants | 17 | 18

3. Primary Outcome: Number of Participants Who do Not Complete the 3-month Post-treatment Follow-up Assessment
Description: A measure of feasibility.
Time Frame: approximately 20-24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HCT Symptoms and Steps | HCT Education
Number analyzed (Participants) | 20 | 20
Participants | 3 | 2

4. Primary Outcome: Acceptability as Measured by the Client Satisfaction Questionnaire (CSQ) 8-item Version
Description: This questionnaire contains 8 items rated from 1=low acceptability to 4=high acceptability; scores are created by utilizing the Likert Scale to sum CSQ answers resulting in a score range from 8 to 32. The intervention is considered acceptable if the mean value for acceptability across all participants is above 80% of max acceptability score (i.e., 25.6).
Time Frame: post-treatment (approximately 7-12 weeks)
Population: Only applicable to the HCT Symptoms and Steps arm. Data not collected on two participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HCT Symptoms and Steps | HCT Education
Number analyzed (Participants) | 18 | 0
units on a scale | 27.89 (3.46) |

5. Secondary Outcome: Change in Physical Disability as Measured by the the Functional Assessment of Cancer Therapy (FACT)
Description: Physical Disability will be assessed using the Functional Assessment of Cancer Therapy 7-item physical well-being scale. Each item is scored 0=not at all to 4=very much as the statement applies to the past 7 days. The full range of the scale is 0 to 28, with a higher score indicating a better outcome.
Time Frame: pre-treatment (baseline), post-treatment (approximately 7-12 weeks)
Population: Participants with data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HCT Symptoms and Steps | HCT Education
Number analyzed (Participants) | 18 | 18
units on a scale | 4.78 (4.91) | 6.94 (6.66)

6. Secondary Outcome: Change in Pain Severity
Description: Pain severity will be assessed with the Brief Pain Inventory (BPI). Patients will rate their "pain right now", "worst", "least" and "average" pain in the last week from 0=no pain to 10=worst pain imaginable. An average of the responses to these items is used to create a single pain severity score.
Time Frame: pre-treatment (baseline), post-treatment (approximately 7-12 weeks).
Population: Participants with data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HCT Symptoms and Steps | HCT Education
Number analyzed (Participants) | 18 | 18
units on a scale | -.79 (2.19) | .02 (1.54)

7. Secondary Outcome: Change in Fatigue
Description: Fatigue will be assessed using the Patient Reported Outcomes Measurement Information System (PROMIS) seven-item Fatigue Scale. For each item, the statement applies to the past 7 days: "never" (1), "rarely" (2), "sometimes" (3), "often" (4), or "always" (5). The summed score is then converted to a T-Score (0-100), where a higher T-Score indicates worse fatigue. 50 indicates the population mean with a standard deviation of 10. 50 and below is considered below average, 50-60 is mild, and 60 or greater is moderate/severe.
Time Frame: pre-treatment (baseline), post-treatment (approximately 7-12 weeks).
Population: Participants with data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HCT Symptoms and Steps | HCT Education
Number analyzed (Participants) | 18 | 18
units on a scale | -2.62 (6.98) | -4.72 (8.73)

8. Secondary Outcome: Change in Physical Activity
Description: Physical Activity will be assessed via step count with a wireless activity tracker (e.g., Fitbit). A distinct value pre and post treatment are reported, no averages were taken across multiple days.
Time Frame: pre-treatment (baseline), post-treatment (approximately 7-12 weeks).
Population: Participants with data collected at both time points.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | HCT Symptoms and Steps | HCT Education
Number analyzed (Participants) | 18 | 18
steps | 1686.35 (3894.57) | 1001.50 (2471.15)

9. Secondary Outcome: Change in Depression
Description: Depression will be assessed using the Hospital Anxiety and Depression Scale (HADS). Each question rated 0-3, totaling 21 points.Total score of 0-7 = normal, 8-10 = borderline abnormal, 11-21 = abnormal.
Time Frame: pre-treatment (baseline), post-treatment (approximately 7-12 weeks)
Population: Participants with data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HCT Symptoms and Steps | HCT Education
Number analyzed (Participants) | 18 | 18
units on a scale | -1.28 (2.49) | -2.72 (5.26)

10. Secondary Outcome: Change in Anxiety.
Description: Anxiety will be assessed using the Hospital Anxiety and Depression Scale (HADS). Each question rated 0-3, totaling 21 points.Total score of 0-7 = normal, 8-10 = borderline abnormal, 11-21 = abnormal.
Time Frame: pre-treatment (baseline), post-treatment (approximately 7-12 weeks)
Population: Participants with data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HCT Symptoms and Steps | HCT Education
Number analyzed (Participants) | 18 | 18
units on a scale | -1.28 (1.96) | -1.22 (2.37)

11. Secondary Outcome: Change in Self-Efficacy
Description: Change in self-efficacy as measured by the Self-Efficacy for Symptom Management scale: 1=not at all confident to 10=totally confident.
Time Frame: pre-treatment (baseline), post-treatment (approximately 7-12 weeks)
Population: Participants with data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HCT Symptoms and Steps | HCT Education
Number analyzed (Participants) | 18 | 18
units on a scale | -.98 (2.47) | .85 (1.52)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from study enrollment through the 3-month follow up, totaling 6 months.
Arm/Group | HCT Symptoms and Steps | HCT Education
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT03859765/Prot_SAP_000.pdf